CLINICAL TRIAL: NCT01202370
Title: A Phase I Study of AR-67 (7-t-butyldimethylsilyl-10-hydroxycamptothecin) Given on Days 1, 4 8, 12 & 15 of an Every 21-day Cycle in Adult Patients With Refractory or Metastatic Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Arno Therapeutics (Industry)
Responsible Party: Principal Investigator, Susanne Arnold, MD, University of Kentucky
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-MULTI-09-MCC
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Solid Malignancies
Keywords: Cancer; Tumors
MeSH Terms: conditions — Neoplasms | interventions — 7-tert-butyldimethylsilyl-10-hydroxycamptothecin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AR-67 (Experimental): Phase 1 study
  Interventions: Drug: 7-t-butyldimethylsilyl-10-hydroxycamptothecin

INTERVENTIONS:
Drug: 7-t-butyldimethylsilyl-10-hydroxycamptothecin — IV Over 1 hour Days 1, 4, 8, 12 & 15 of a 21 day cycle (7.5 mg/m^2).
  Other Names: AR-67

SUMMARY:
Camptothecins are a potent class of anticancer drugs that inhibit DNA Topoisomerase I. While seen strictly as cytotoxic compounds, camptothecins are actually also targeted agents, inhibiting DNA-Topoisomerase I (Topo I) cleavable complex. First and second generation cogeners are hampered by a labile α-hydroxy-δ-lactone pharmacophore, which hydrolyzes to yield the inactive carboxylate form of the drug. AR-67 (7-t-butyldimethylsilyl-10-hydroxycamptothecin) is a third generation analog engineered to be stable in blood and highly potent. Its enhanced stability results from two factors: (1) AR-67 is highly lipophilic, partitioning into lipid bilayers, thus protecting it from hydrolysis in the aqueous milieu of the bloodstream, and (2) the 10-hydroxy functionality of the drug effectively ablates the high affinity interactions of the carboxylate drug form with albumin, which has been previously shown to diminish the levels of the active lactone species in the circulation. In a recently completed phase I trial, AR-67 showed over 85% lactone stability at all time points studied, and was well-tolerated with grade 4 thrombocytopenia, neutropenic fever and grade 3 fatigue as dose limiting toxicities. The MTD was established at 7.5 mg/m2/day in a daily times five of a 21 day cycle. Preclinical data indicates that AR-67 may concentrate in tumors for a prolonged period of time, compared to plasma clearance of the drug, a phenomenon which has the potential to improve efficacy and decrease toxicity of this compound. What is not known is the optimal dose and schedule of AR-67 needed to produce high tumor penetration, and modest systemic exposure. This pilot proposal seeks to study AR-67 in a novel dosing schedule and to evaluate the feasibility of performing tumor biopsies to determine the tumor half-life of AR-67 in humans. By using multiple tumor biopsies, as a means to document penetration of tumor tissue by AR-67, and compare that to plasma clearance of the drug, the investigators will establish direct pharmacokinetic evidence that AR-67 "hits the target". The investigators propose that a rigorous evaluation of drug penetration into the tumor should be considered, in addition to the MTD, when determining dose of new experimental compounds. Dose-tumor concentration relationships should be established early in the course of clinical development to provide data for rational selection of the phase-II dose. This pilot study will provide important preliminary data to establish the feasibility of this approach for future study. If successful, tumor half life will be used to develop an optimal biologic dose in a phase I trial using this schedule of AR-67. Optimal biologic dosing could become a new standard for dose escalation studies with this compound and other cytotoxic drugs that have specific biologic targets in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or greater and have a histologically or cytologically proven solid malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Patients who have recurred after previous surgery and/or radiation may participate in this trial, although no restriction is placed on the number of prior therapies. Patients must be willing and able to have two core-needle biopsies of their tumor to participate in this trial.
* Patients with known brain metastases are eligible for this clinical trial if their disease has been treated and they are clinically stable (based on the assessment of their treating physician) and documented by a stable or improved pretreatment CT or MRI scan of the brain to evaluate for CNS disease within 28 days prior to registration.
* Patients may have measurable OR non-measurable disease documented by CT, MRI, X-ray or nuclear exam (FDG-PET). All disease must be assessed within 28 days prior to registration. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of measurable disease.
* Patients must have progressed after at least one prior chemotherapy and not be candidates for salvage surgery. Prior biologic therapy or prior radiation is permitted; however, at least two weeks must have elapsed since the completion of prior therapy and patients must have recovered from all associated toxicities (due to prior therapy) at the time of registration.
* At least three weeks must have elapsed since surgery (thoracic or other major surgeries) and patients must have recovered from all associated toxicities at the time of registration.
* Patients must have acceptable organ and marrow function documented within seven days of registration and as defined below:

  * Leukocytes >3,000/mcL
  * Absolute neutrophil count >1,500/mcL
  * Platelets >100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional ULN
  * Creatinine within normal institutional limits, OR
  * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of <2.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 3 years.
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including fetal death from the chemotherapeutic agents. In order to participate in this trial, women / men of reproductive potential must agree to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Women of childbearing potential must have a negative serum pregnancy test documented within seven days of registration.
* Patients must be informed of the investigational nature of this study and must sign and provide a written informed consent in accordance with institutional and federal guidelines.
* Patients must have a life expectancy of greater than 12 weeks.
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of AR-67 will be determined following review of their case by the Principal Investigator. Efforts should be made to switch patients taking drugs that are strong inducers of the enzyme CYP3A4 including anticonvulsants (i.e., phenytoin, phenobarbital, carbamazepine, or primidone) and rifampin OR strong inhibitors of CYP3A4 (clarithromycin, itraconazole, and ketoconazole) to other appropriate medications

Exclusion Criteria:

* Patients must not have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of ≥ Grade 3 allergic reactions attributed to compounds of similar chemical or biologic composition to AR-67 (i.e. camptothecins such as irinotecan, topotecan or others of this class of pharmaceuticals).
* Patients with prior anaphylactic injection reaction of > Grade 3 to paclitaxel or any other product formulated with Cremophor.
* Pregnant women are excluded from this study because AR-67 is a camptothecin with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AR-67, breastfeeding should be discontinued if the mother is treated with AR-67.
* HIV-associated symptoms may preclude accurate assessment of toxicity or response to the treatment and because the primary endpoint of this Phase I trial is toxicity, patients with HIV disease will be ineligible for participation. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AR-67. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and are ineligible for enrollment on this study.
* Subjects with leukemia or primary brain tumors are excluded from this study.
* Subjects may not receive any of the following medications two weeks prior to, during or two weeks after initiation of AR-67: aprepitant, atazanavir, bacillus of Calmette and Guerin vaccine, carbamazepine, citalopram, ketoconazole, intraconazole, measles virus vaccine, mumps virus vaccine, phenobarbital, phenytoin, poliovirus vaccine, rifabutin, rifampin, rotavirus vaccine, rubella virus vaccine, smallpox vaccine, St John's wort, typhoid vaccine, varicella virus vaccine or yellow fever vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of obtaining two serial tumor biopsies and plasma pharmacokinetics for the determination of AR-67 half life in tumor and plasma during day 1 of AR-67 treatment given on days 1, 4, 8, 12 and 15 of an every 21-day cycle. | Cycle 1 days 1 and 2

SECONDARY OUTCOMES:
Toxicities | Days 1, 4, 8, 12 and 15 of an every 21-day cycle
  To document all toxicities of AR-67 after intravenous (IV) administration on days 1, 4, 8, 12 and 15 of an every 21-day cycle to adults with recurrent or refractory solid tumors in which standard therapies are not effective.
Feasibility for testing topoisomerase-I and γ-H2AX in tumor tissue | Cycle 1 days 1 and 2
  To determine the feasibility for testing the expression of topoisomerase-I and γ-H2AX in tumor tissue biopsies using immunohistochemical techniques and western blot assays.
Efficacy | Days 1, 4 , 8, 12 and 15 of a 21 day cycle
  To collect efficacy data for these subjects using radiographic assessment of tumor response by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Arnold, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States